CLINICAL TRIAL: NCT05479578
Title: A Phase I Study of Oral Metronomic Dosing of Oral Cyclophosphamide with Dexamethasone for Metastatic Castration Resistant Prostate Cancer
Brief Title: Cyclophosphamide and Dexamethasone for the Treatment of Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rashmi Verma, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Rashmi Verma, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#301; NCI-2022-05133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#301 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-07-29 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer American Joint Committee on Cancer (AJCC) V8
MeSH Terms: interventions — Cyclophosphamide; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cyclophosphamide, dexamethasone) (Experimental): Patients receive cyclophosphamide PO QD and dexamethasone PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex

SUMMARY:
This phase I trial tests the safety and side effects of cyclophosphamide given together with dexamethasone in treating patients with castration resistant prostate cancer that has spread to other places in the body (metastatic). Chemotherapy drugs, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving low doses of cyclophosphamide daily may reduce side effects. Dexamethasone is a corticosteroid drug that is used to treat some of the problems caused by chemotherapy treatment. The combination of cyclophosphamide and dexamethasone may work better in treating patients with castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate the feasibility of using the combination of oral metronomic cyclophosphamide and oral dexamethasone for treatment of men with metastatic castration -resistant prostate Cancer (mCRPC) who have progressed on 2 or more prior treatments. II. To assess the safety of cyclophosphamide + dexamethasone in men with mCRPC who have progressed on 2 or more prior treatments. SECONDARY OBJECTIVE:I. To evaluate prostate specific antigen (PSA) response and progression free survival and time to event outcome in participants with mCRPC treated with cyclophosphamide and dexamethasone. EXPLORATORY OBJECTIVE: I. To analyze serial blood samples for PSA monitoring and tumor tissue for pRb (encoded by the RB1 gene) and p53 (encoded by the TP53 gene) mutations. OUTLINE: Patients receive cyclophosphamide orally (PO) once daily (QD) and dexamethasone PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements
* Adults >= 18 years of age at time of consent
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 or 2
* Life expectancy >= 3 months
* Histologically or cytologically confirmed prostate adenocarcinoma
* Metastatic status defined as at least 1 documented metastatic lesion on a bone scan, a computed tomography (computed tomography [CT] or CT/ positron emission tomography [PET]) scan, or a magnetic resonance imaging (MRI) scan
* Must have less than 50 ng/dL testosterone
* Must have demonstrated disease progression after treatment with 2 or more prior lines of therapies for castration resistant prostate cancer (CRPC), including one second generation androgen targeted agent (such as abiraterone or enzalutamide).
* PSA defined progression after most recent directed therapy. Progression is defined as PSA increase >= 25% of baseline or absolute increase of >= 2 ug/L on two PSA measurements at least 7 days apart
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 8 g/dL
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) range
* Aspartate aminotransferase (AST) and alanine transaminase (ALT) levels =< 2.5 × ULN or AST and ALT levels =< 5 x ULN (for participants with documented metastatic disease to the liver)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (for participants on anticoagulation they must be receiving a stable dose for at least 1 week prior to first treatment)
* Creatinine clearance > 30 mL/min by Cockcroft-Gault formula
* Participants with BRCA1/2 or homologous recombination (HR) deoxyribonucleic acid (DNA) repair mutations, and/ or microsatellite instability (MSI) must have received prior treatment (e.g., PARP [poly adenosine diphosphate-ribose polymerase] inhibitors or other agents) for BReast CAncer gene (BRCA)/ homologous recombination (HR) DNA repair mutation and/ or MSI
* Participants with known active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is < 100 IU/mL prior to first dose of trial treatment. Participants with treated or untreated hepatitis C virus (HCV) are allowed.
* Male participants who agree to use highly effective method of birth control with their partner (e.g., implants, injectables, birth control pills with two hormones, intrauterine devices [IUDs], complete abstinence or sterilized partner, and female sterilization) and a barrier method (e.g., condoms, vaginal ring, sponge, etc.) during the period of therapy and for 90 days after the last dose of study drug

Exclusion Criteria:

* Any condition that would prohibit the understanding or rendering of informed consent
* A history of any other active malignancy with progression and requiring treatment/intervention, with the exception of cutaneous malignancies such as basal cell carcinoma, squamous cell carcinoma, melanoma, or the type of malignancy being studied in this protocol
* Participants with urinary outflow obstruction that has not been treated or managed with either indwelling catheter or self-catheterization
* Severe untreated infection that in the opinion of the investigator would interfere with participant safety or compliance on trial within 28 days prior to enrollment
* Any condition, including concomitant disease, additional malignancies, laboratory abnormalities, or psychiatric illness, that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial
* Use of systemic therapy for the treatment of prostate adenocarcinoma within 2 weeks of initiating study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Treatment initiation through treatment completion, an average of up to 4 years
  Feasibility, defined as >= 80% of participants completing treatment, and safety as defined by Grade 3 or higher adverse events (AEs) observed per National Cancer Institute (NCI) Common Terminology Criteriafor Adverse Events (CTCAE 5.0) criteria
Incidence of adverse events | Treatment initiation through treatment completion, an average of up to 4 years
  Number of participants experiencing adverse events (AEs), both non treatment related and treatment related, classified by severity and graded.

SECONDARY OUTCOMES:
Total prostate-specific antigen (PSA) response rate | From date of treatment initiation through PSA response (as defined by Prostate Cancer Working Group 2 [PCWG2]), an average of up to 4 years
  Defined as a decline in PSA of 50% or greater, confirmed evaluation every 28 days with no evidence of clinical progression or disease progression on imaging, consistent with previous definitions by the Prostate Cancer Working Group 2 (PCWG2). The PSA response rate will be estimated along with an exact 95% confidence interval. Kaplan-Meier analysis will be used to depict time-to-event outcomes graphically and estimate medians with 95% confidence intervals.
Time to no longer clinical benefit (NLCB) | Treatment initiation through treatment completion, an average of up to 4 years
Time to prostate-specific antigen (PSA) progression | From date of treatment initiation to PSA progression (as defined by Prostate Cancer Working Group 2 [PCWG2]), an average of up to 4 years
Time to radiographic progression free survival (rPFS) | From date of treatment initiation to radiographic progression (as defined by Prostate Cancer Working Group 2 [PCWG2]) or date of death from any cause, whichever came first, an average of up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Verma, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States